CLINICAL TRIAL: NCT05719519
Title: Change in Gingival Volume and Quality of Life Due to Initial Periodontal Therapy in Smokers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rijeka (Other)
Responsible Party: Principal Investigator, Aleksandar Pupovac, Assistant, Department of periodontology, University of Rijeka
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 08-21
Record Dates: First submitted 2023-01-25; First posted 2023-02-09 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Periodontitis
Keywords: 3D imaging; gingiva; nonsurgical periodontal debridement; periodontitis; quality of life; smoking
MeSH Terms: conditions — Periodontitis; Smoking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smokers (Other)
  Interventions: Procedure: Initial periodontal therapy and 3D intraoral scanning
- Non smokers (Experimental)
  Interventions: Procedure: Initial periodontal therapy and 3D intraoral scanning

INTERVENTIONS:
Procedure: Initial periodontal therapy and 3D intraoral scanning — Initial periodontal therapy using GBT ( guided biofilm therapy) principle and 3D intraoral scanning

SUMMARY:
The aim of this study is to compare the dimensional changes of the gingiva due to initial periodontal therapy in non-smokers and cigarette smokers and to compare the oral health related quality of life of non-smokers and cigarette smokers with periodontitis before and after initial periodontal therapy. Changes in gingival volume are expected to be greater in non-smokers than in cigarette smokers. It is expected that the quality of life will be better after therapy in both groups, with better results in the non-smoking group.

60 subjects with periodontitis will be included in the study 30 non-smokers and 30 cigarette smokers. All subjects will fill out a quality of life questionnaire which will be validated before the onset of this research. This will be followed by clinical periodontal examination. After examination, the upper and lower jaw will be scanned using an intraoral scanner and initial periodontal therapy will be performed. After 8 weeks, subjects will fill out the quality of life questionnaire again, measurement of periodontal indices and scanning will be performed. The digital scans wll be superimposed, and the dimensional changes of the gingiva will be quantified and compared between the two groups. By using 3D technology, it will be possible to objectively quantify tissue changes and monitor the course of the disease. A 3D comparison between non-smokers and cigarette smokers will provide a new perspective on the relationship between smoking and periodontitis. Furthermore, it will be demonstrated to what extent smoking affects the quality of life of patients with periodontitis and the results of non-surgical therapy.

ELIGIBILITY:
Inclusion Criteria:

* periodontitis
* cigarette smokers
* non smokers

Exclusion Criteria:

* previous periodontal treatment
* pregnancy
* minors
* antibiotic therapy in the last 6 months
* patients with ortho appliances
* patients using drugs that affect gingival volume
* immunosuppressive therapy
* systemic conditions that affects periodontal tissues and therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Volume changes | 24 months
  soft tissue volume changes after therapy ( mm3)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pupovac A, Kuis D, Miskovic I, Spalj S, Zhurov A, Prpic J. A New Method for Volumetric Analysis of Soft-Tissue Changes Using Three-Dimensional Imaging in Patients With Periodontitis. J Clin Periodontol. 2025 Jun;52(6):888-897. doi: 10.1111/jcpe.14118. Epub 2025 Apr 15. PMID 40234017